CLINICAL TRIAL: NCT05961527
Title: An Open-Label Feasibility and Safety Study of MDMA-Assisted Group Therapy for the Treatment of Posttraumatic Stress Disorder in Veterans
Brief Title: Group MDMA-therapy for Veterans With PTSD
Acronym: Group-MVP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Portland VA Research Foundation, Inc (Other)
Collaborators: Steven & Alexandra Cohen Foundation (Other)
Responsible Party: Principal Investigator, Christopher Stauffer, Associate Professor of Psychiatry, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02
Record Dates: First submitted 2023-07-17; First posted 2023-07-27 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: PTSD
Keywords: MDMA; PTSD; Veterans; Group Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Psychotherapy, Group

STUDY DESIGN:
Intervention Model Description: Open-label study examining safety and feasibility of MDMA-assisted group therapy
Masking Description: Independent raters for the primary clinical outcome will be blinded to study design and timepoint.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- MDMA-assisted group therapy (Experimental): Four Preparatory Sessions, two MDMA Sessions, and four Integrative Sessions following each MDMA Session.
  Interventions: Drug: MDMA; Behavioral: Group Therapy

INTERVENTIONS:
Drug: MDMA — Initial dose of 120 mg MDMA HCL and optional supplemental dose of 60 mg MDMA HCL at 1.5 to 2 hours after first dose
  Other Names: 3,4-methylenedioxymethamphetamine
Behavioral: Group Therapy — Standardized group psychotherapy performed by therapist team in combination with non-directive MDMA therapy

SUMMARY:
This Phase 2a, open-label, non-randomized, 3-cohort study assesses the feasibility and safety of MDMA-assisted group therapy for the treatment of PTSD in veterans. The study will be conducted in up to N=18 participants, recruited in three cohorts of six participants each and receive therapy sessions throughout their participation in these group cohorts.

DETAILED DESCRIPTION:
To assess the feasibility and safety of MDMA-assisted group therapy for participants with at least moderate PTSD, the sponsor-investigator is conducting a phase 2, open-label, non-randomized, 3-cohort study. This novel treatment package consists of two once-monthly open-label MDMA Sessions combined with non-drug preparatory and integrative therapy administered in both individual and group sessions. The Primary Clinical Outcome measure, the Clinician Administered PTSD Scale (CAPS-5), evaluates changes in PTSD symptom severity and is assessed by a blinded centralized Independent Rater (IR) pool. The therapeutic approach will combine manualized MDMA-assisted therapy for PTSD with group therapy components.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years old.
* Are a U.S. Military Veteran
* Are fluent in speaking and reading the predominantly used or recognized language of the study site.
* Are able to swallow pills.
* Agree to have study visits recorded, including MDMA Sessions, outcome assessments, and non-drug psychotherapy sessions.
* Must provide a contact who is willing and able to be reached by the investigators in the event of a participant becoming suicidal or unreachable.
* Must agree to inform the investigators within 48 hours of any medical conditions and procedures.
* If able to become pregnant, must have a negative pregnancy test at study entry and prior to each Experimental Session, and must agree to use adequate contraception through 10 days after the last Experimental Session.
* Must not participate in any other interventional clinical trials during the duration of the study.
* Must commit to medication dosing, therapy, and study procedures.
* Have a current PTSD diagnosis at the time of screening.

Exclusion Criteria:

* Are not able to give adequate informed consent.
* Have uncontrolled hypertension.
* Have a marked baseline QTcF interval >450 milliseconds [ms] demonstrated on repeated ECG assessments.
* Have a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
* Have evidence or history of significant medical disorders.
* Have symptomatic liver or biliary disease.
* Have history of hyponatremia or hyperthermia.
* Weigh less than 48 kilograms (kg).
* Are pregnant or nursing, or are able to become pregnant and are not practicing an effective means of birth control.
* Are abusing illegal drugs or alcohol.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Change in CAPS-5 Total Severity Score | Baseline - 3 months from first Experimental Session
  The CAPS-5 is a semi-structured interview that assesses index history of DSM-5-defined traumatic event exposure, including the most distressing event, time since exposure, to produce a diagnostic score (presence vs. absence) and a PTSD Total Severity score. The CAPS-5 rates intrusion symptoms (intrusive thoughts or memories), avoidance, cognitive and mood symptoms, arousal and reactivity symptoms, duration and degree of distress and dissociation. The total severity score is a sum of symptom frequency and intensity scores for the subscales B (re-experiencing), C (avoidance) and D (hypervigilance) and ranges from 0 to 136, with higher scores indicating greater severity of PTSD symptoms.

SECONDARY OUTCOMES:
Change in Sheehan Disability Scale (SDS) | Baseline - 3 months from first Experimental Session
  Sheehan Disability Scale (SDS) total score, a measure of clinician-rated functional impairment. The first three items indicate degree of impairment in the domains of work/school, social life, and home life, with response options based on an eleven-point scale (0=not at all to 10=extremely), and five verbal tags (not at all, mildly, moderately, markedly, extremely). The remaining two items assess Days Lost and Days Unproductive during the reporting period.

CONTACTS AND LOCATIONS:
Locations (1):
- Portland-Vancouver VA, Vancouver, Washington, United States

IPD SHARING:
Plan to Share IPD: No